CLINICAL TRIAL: NCT00452413
Title: A Phase 1/2 Trial of Enzastaurin and Erlotinib in Patients With Advanced Solid Tumors and Non-Small Cell Lung Cancer (NSCLC) After Prior Chemotherapy
Brief Title: A Study of Enzastaurin and Erlotinib in Participants With Solid Tumors and Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11183; H6Q-MC-S030 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Non-Small Cell Lung Cancer; Malignant Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — enzastaurin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin and erlotinib combination therapy (Experimental): Enzastaurin:
  * Phase 1, Dose Level 1: 500 milligram (mg) oral loading dose Day 1, 250 mg oral, daily Day 2-28, 28-day cycle until disease progression
  * Phase 1, Dose Level 2: 1125 mg oral loading dose Day 1, 500 mg oral, daily until disease progression
  * Phase 2: Dose determined from Phase 1, oral, daily, 28-day cycles until disease progression
  Erlotinib:
  • 150 mg, oral, daily, 28-day cycles until disease progression
  Interventions: Drug: enzastaurin; Drug: erlotinib

INTERVENTIONS:
Drug: enzastaurin — Administered orally
  Other Names: LY317615
Drug: erlotinib — Administered orally

SUMMARY:
Phase I: A study to see what doses of Enzastaurin and Erlotinib are best tolerated by participants with solid tumor cancer.

Phase II: A study to see how long participants with non-small cell lung cancer (NSCLC) treated with Enzastaurin and Erlotinib live.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1: Any incurable solid malignancy, with no more than 3 prior systemic treatment regimens.

   Phase 2: Histologic diagnosis of advanced NSCLC, Stage IIIB with malignant pleural effusion or Stage IV per American Joint Committee on Cancer Staging Criteria for NSCLC. Participants must have failed 1 or 2 prior systemic treatment regimen(s).
2. Performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Scale
3. Prior chemotherapy must be completed at least 2 weeks prior to study enrollment, and the participant must have recovered from acute toxic effects (except alopecia) prior to enrollment.
4. Prior radiotherapy is allowed to <25% of the bone marrow. Prior radiotherapy must be completed at least 2 weeks before study enrollment, and the participant must have recovered from acute toxic effects (except alopecia) prior to enrollment.
5. Non-measurable or measurable disease as defined by Response Evaluation Criteria in Solid Tumors [RECIST, version (v) 1.0].

Exclusion Criteria:

Participants who

1. Are unable to swallow tablets.
2. Unable to discontinue use of carbamazepine, phenobarbital, and phenytoin.
3. Have previously been treated with an epidermal growth factor receptor (EGFR) inhibitor, including erlotinib.
4. Are receiving concurrent administration of any other antitumor therapy.
5. Have received treatment within the last 30 days with a drug (not including study drug) that has not received regulatory approval for any indication at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas

REFERENCES:
- [Derived] Padda SK, Krupitskaya Y, Chhatwani L, Fisher GA, Colevas AD, San Pedro-Salcedo M, Decker R, Latz JE, Wakelee HA. A phase I dose-escalation and pharmacokinetic study of enzastaurin and erlotinib in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2012 Apr;69(4):1013-20. doi: 10.1007/s00280-011-1792-8. Epub 2011 Dec 11. PMID 22160298
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included 2 phases: Phase 1, a dose-escalation phase (employing a standard "3 + 3" design with dose escalation to Dose Level 2 based upon observed toxicity) and Phase 2, a dose-confirmation phase.
Groups:
- Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg): Enzastaurin: 500 milligram (mg) enzastaurin loading dose [250 mg twice daily (BID)] administered orally on Day 1 of a 28-day cycle. Day 2 through Day 28, 250 mg dose administered once daily (QD).
  Erlotinib: 150 mg dose of erlotinib administered orally QD.
  Treatment continued until disease progression, unacceptable toxicity, or study withdrawal criteria were met.
- Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg): Enzastaurin: 1125 mg enzastaurin loading dose [375 mg 3 times daily (TID)] administered orally on Day 1 of a 28-day cycle. Day 2 through Day 28, 500 mg dose administered QD.
  Erlotinib: 150 mg dose of erlotinib administered orally QD.
  Treatment continued until disease progression, unacceptable toxicity, or study withdrawal criteria were met.
- Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg): Enzastaurin: 1125 mg enzastaurin loading dose (375 mg TID) administered orally on Day 1 of a 28-day cycle. Day 2 through Day 28, 500 mg total daily dose administered orally using either a BID or QD schedule.
  Erlotinib: 150 mg dose of erlotinib administered orally QD.
  Treatment continued until disease progression, unacceptable toxicity, or study withdrawal criteria were met.
Period: Overall Study
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg) | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Started | 4 | 12 | 49
Received at Least 1 Dose of Study Drug | 4 | 12 | 49
Completed | 0 | 0 | 0
Not Completed | 4 | 12 | 49
Not completed — Progressive Disease | 4 | 11 | 30
Not completed — Withdrawal by Subject | 0 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Death due to study disease | 0 | 0 | 2
Not completed — Death due to adverse event (AE) | 0 | 0 | 1
Not completed — On treatment | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Enrolled participants who received at least 1 dose of study drug (either enzastaurin or erlotinib).
Groups:
- Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg): Enzastaurin: 500 mg enzastaurin loading dose (250 mg BID) administered orally on Day 1 of a 28-day cycle. Day 2 through Day 28, 250 mg dose administered QD.
  Erlotinib: 150 mg dose of erlotinib administered orally QD.
  Treatment continued until disease progression, unacceptable toxicity, or study withdrawal criteria were met.
- Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg): Enzastaurin: 1125 mg enzastaurin loading dose (375 mg TID) administered orally on Day 1 of a 28-day cycle. Day 2 through Day 28, 500 mg dose administered QD.
  Erlotinib: 150 mg dose of erlotinib administered orally QD.
  Treatment continued until disease progression, unacceptable toxicity, or study withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg) | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg) | Total
Number analyzed (Participants) | 4 | 12 | 49 | 65
Age, Continuous [Median (Full Range); unit: years] | 74.0 (10.5) [60 to 83] | 62.5 (8.45) [46 to 75] | 67.0 (9.19) [42 to 83] | 66.0 (NA) [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 20 | 33
  Male | 0 | 3 | 29 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 8 | 38 | 49
  Hispanic | 0 | 1 | 1 | 2
  East Asian | 1 | 3 | 7 | 11
  African | 0 | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 12 | 49 | 65
Stage of Disease at Initial Diagnosis [Count of Participants; unit: Participants] — Classification based on American Joint Committee on Cancer (AJCC) Staging System for lung cancer (sixth edition, 2002). Disease stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIB is a locally advanced cancer that has spread to nearby tissues or far away lymph nodes, or has fluid, containing cancer cells, built up between the layers lining the lungs.
  Participants
    Stage IIIB | 0 | 1 | 6 | 7
    Stage IV | 4 | 11 | 43 | 58

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose for Enzastaurin Plus Erlotinib Combination Therapy (Assess the Tolerated Dose of the Combination Erlotinib and Enzastaurin)
Description: The recommended Phase 2 daily dose level was to be either 1 dose level below that in which 2 of 6 participants experienced dose-limiting toxicities (DLTs) in Phase 1 or the full doses of both enzastaurin and erlotinib (Phase 1, Dose Level 2) in the event that no more than 1 DLT occurred at the highest dose level (Dose Level 2). DLTs were defined as any of the following events during Phase 1, Cycle 1 that were considered by the investigator to be attributable to enzastaurin or the combination of enzastaurin with erlotinib: Grade 4 hematologic events; Grade 3 or 4 nonhematologic events except toxicities explained by a coexisting condition such as glucose disturbances in a diabetic or electrolyte imbalances from diarrhea or vomiting, and toxicities of nausea, vomiting, diarrhea, or skin rash that were tolerable with appropriate treatment.
Time Frame: Phase 1: Predose through end of Cycle 1 (28 days/cycle)
Population: Participants enrolled in Phase 1 who received at least 1 dose of study drug (either enzastaurin or erlotinib).
Measure: Number; unit: milligrams per day (mg/day)
Groups:
- Phase 1, Dose 1 and 2 (Enzastaurin and Erlotinib): Enzastaurin: Either 500 mg or 1125 mg enzastaurin loading dose administered orally on Day 1 of a 28-day cycle. Day 2 through Day 28, either 250 mg or 500 mg dose administered QD.
  Erlotinib: 150 mg dose of erlotinib administered orally QD.
  Treatment continued until disease progression, unacceptable toxicity, or study withdrawal criteria were met.
Arm/Group | Phase 1, Dose 1 and 2 (Enzastaurin and Erlotinib)
Number analyzed (Participants) | 16
milligrams per day (mg/day)
  Enzastaurin | 500
  Erlotinib | 150

2. Primary Outcome: Phase 2: Progression-Free Survival (PFS) With the Enzastaurin Plus Erlotinib Combination Regimen
Description: PFS was defined as the time from the date of study enrollment (baseline) to the first date of progressive disease (PD) (either objectively determined or clinical progression) or death from any cause. PD was defined by Response Evaluation Criteria in Solid Tumors [RECIST, version (v) 1.0] as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. For participants not known to have died as of the data cut-off date and who did not have PD, PFS was censored at the date of the last visit with adequate assessment. For participants who received subsequent anticancer therapy (after discontinuation from study treatment) prior to disease progression or death, PFS was censored at the date of last visit with adequate assessment prior to the initiation of post discontinuation anticancer therapy.
Time Frame: Phase 2: Baseline to measured PD (up to 20 months)
Population: Participants enrolled in Phase 2 who received at least 1 dose of study drug (either enzastaurin or erlotinib). Eight participants were censored.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 41
months | 1.7 [1.5 to NA] — The measure of dispersion was a 1-sided confidence interval at the significance level of 0.10.

3. Secondary Outcome: Phase I: Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs) (Safety and AE Profile for Enzastaurin/Erlotinib Combination)
Description: A TEAE is any untoward medical occurrence that either occurred or worsened any time after treatment baseline, which did not necessarily have a causal relationship with this treatment. A summary of serious and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Phase 1: First dose through 30 days post last dose (up to 14 Cycles, 28 days/cycle)
Population: Participants enrolled in Phase 1 who received at least 1 dose of study drug (either enzastaurin or erlotinib).
Measure: Number; unit: Participants
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 4 | 12
Participants | 4 | 12

4. Secondary Outcome: Phase I: Pharmacokinetic (PK) Interactions Between Enzastaurin and Erlotinib: Apparent Oral Clearance of Erlotinib Under Steady State Conditions During Multiple Dosing (CLss/F)
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL obtained after an oral dose (apparent oral CL) is influenced by the fraction of the dose absorbed (F). Drug CL is a quantitative measure of the rate at which a drug substance is removed from the blood. Apparent oral CL of erlotinib over 10 hours at steady state (ss) on Day 22 was calculated.
Time Frame: Phase 1: Cycle 1, Day 22 [predose, 2 hours (h), 4 h, 6 h, 10 h postdose]
Population: Participants enrolled in Phase 1 who received at least 1 dose of study drug (enzastaurin or erlotinib) and had adequate sample data to estimate CLss/F of erlotinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 3 | 11
Liters per hour (L/h) | 6.07 (19) | 5.75 (45)

5. Secondary Outcome: Phase I: PK Interactions Between Enzastaurin and Erlotinib: Maximum Observed Plasma Concentration at Steady State (Cmax,ss)
Description: Maximum observed plasma concentration at steady state (Cmax,ss) of enzastaurin, its active metabolite (LSN326020) and total analyte were reported.
Time Frame: Phase 1: Cycle 1, Day 22 (predose, 2 h, 4 h, 6 h, 8 h postdose)
Population: Participants enrolled in Phase 1 who received at least 1 dose of study drug (enzastaurin or erlotinib) and had adequate sample data to estimate Cmax,ss of enzastaurin, its active metabolite and total analyte.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 3 | 12
nanomoles per liter (nmol/L)
  Enzastaurin | 618 (709) | 1600 (57)
  LSN326020 | 431 (806) | 980 (41)
  Total Analyte | 978 (797) | 2620 (44)

6. Secondary Outcome: Phase I: PK Interactions Between Enzastaurin and Erlotinib: Area Under the Plasma Concentration Time Curve at Steady State [AUC(Tau,ss)]
Description: Area under the plasma concentration time curve AUC(Tau,ss) of enzastaurin, its active metabolite (LSN326020) and total analyte were reported.
Time Frame: Phase 1, Cycle 1, Day 22 (predose, 2 h, 4 h, 6 h, and 8 h postdose)
Population: Participants enrolled in Phase 1 who received at least 1 dose of study drug (enzastaurin or erlotinib) and had adequate sample data to estimate AUC(Tau,ss) of enzastaurin, its active metabolite, and total analyte.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hours per liter (nmol*h/L)
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 3 | 12
nanomoles*hours per liter (nmol*h/L)
  Enzastaurin | 6590 (412) | 18000 (71)
  LSN326020 | 7100 (890) | 18000 (44)
  Total Analyte | 14000 (598) | 37100 (51)

7. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of study enrollment (baseline) to the date of death from any cause. For participants not known to have died as of the data cutoff date, OS was censored at the last contact date (last contact for participants in post discontinuation was equal to the last known alive date in mortality status).
Time Frame: Phase 2: Baseline to date of death from any cause (up to 23 months)
Population: Participants enrolled in Phase 2 who received at least 1 dose of study drug (either enzastaurin or erlotinib). Eighteen participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 31
months | 8.3 [5.3 to 14.3]

8. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response: time from first objective assessment of complete response (CR) or partial response (PR) to first observation of PD. Using RECIST v1.0 criteria, CR was the disappearance of all target lesions; PR was either a ≥30% decrease in sum of LD of target lesions or a complete disappearance of target lesions, with persistence (but not worsening) of ≥1 nontarget lesion; PD was a ≥20% increase in sum of LD of target lesions, taking as references the smallest sum LD recorded since treatment started or the appearance of ≥1 new lesion. For responding participants not known to have died and who did not have PD, duration of response was censored at date of the last visit with adequate assessment. For responding participants who received subsequent anticancer therapy (after discontinuation from study treatment) prior to PD, duration of response was censored at the date of last visit with adequate assessment prior to the initiation of post discontinuation anticancer therapy.
Time Frame: Phase 2: Date of first response to date of PD (up to 18 months)
Population: Participants enrolled in Phase 2 who received at least 1 dose of study drug (either enzastaurin or erlotinib) and had a CR or PR response. Two participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 3
months | 8.7 [7.5 to NA] — The upper 95% confidence interval was not estimable because an insufficient number of participants reached the event at the final time point for assessment.

9. Secondary Outcome: Phase 2: Percentage of Participants With Tumor Response
Description: Tumor response was defined using RECIST, v1.0 criteria. CR was the disappearance of all target lesions; PR was either a ≥30% decrease in sum of LD of target lesions or a complete disappearance of target lesions, with persistence (but not worsening) of ≥1 nontarget lesion. PD was a ≥20% increase in sum of LD of target lesions, taking as references the smallest sum LD recorded since treatment started or the appearance of ≥1 new lesion. Stable Disease (SD) was defined as small changes that did not meet the above criteria. Percentage of participants with tumor response=[(number of participants with a CR, PR, SD, PD, and unknown response)/(total number of participants assessed)]*100.
Time Frame: Phase 2: Baseline to date of PD (up to 18 months)
Population: Participants enrolled in Phase 2 who received at least 1 dose of study drug (either enzastaurin or erlotinib).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 49
percentage of participants
  CR | 0 [0 to 7.3]
  PR | 10.2 [3.4 to 22.2]
  SD | 20.4 [10.2 to 34.3]
  PD | 42.9 [28.8 to 57.8]
  Unknown | 26.5 [14.9 to 41.1]

10. Secondary Outcome: Phase 2: Number of Participants Who Experienced TEAEs (Safety and AE Profile)
Description: as for outcome 3
Time Frame: Phase 2: Baseline through 30 days post last dose (up to 24 Cycles, 28 days/cycle)
Population: Participants enrolled in Phase 2 who received at least 1 dose of study drug (either enzastaurin or erlotinib).
Measure: Number; unit: participants
Arm/Group | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Number analyzed (Participants) | 49
participants | 48

ADVERSE EVENTS:
Arm/Group | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg) | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg)
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/12 | 18/49
Other Adverse Events (participants affected / at risk) | 4/4 | 12/12 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) (N=4) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg) (N=12) | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg) (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug interaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1, Dose 1 (Enzastaurin 250 mg, Erlotinib 150 mg) (N=4) | Phase 1, Dose 2 (Enzastaurin 500 mg, Erlotinib 150 mg) (N=12) | Phase 2 (Enzastaurin 500 mg, Erlotinib 150 mg) (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Nucleated red cells (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 2 (5)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 2 (2) | 4 (4)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelash thickening (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Growth of eyelashes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 11 (13) | 36 (54)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 7 (8) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 8 (9) | 21 (23)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oral papule (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (7) | 12 (12)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 3 (3) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 9 (10) | 21 (26)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 3 (3)
Pain (General disorders) | 0 (0) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (6)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 5 (5)
Vaginal abscess (Infections and infestations) | 0 (0) | 0/9 (0) | 1/20 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferase decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Band neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 4 (6)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood lactate dehydrogenase decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood methaemoglobin present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Neutrophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prealbumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Romberg test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 9 (10)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (8) | 19 (24)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 9 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (4)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 6 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 6 (6)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 7 (7)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 3 (3) | 9 (9) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1/3 (1) | 0/29 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1/3 (1) | 0/29 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0/9 (0) | 1/20 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1/9 (1) | 0/20 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 14 (18)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 12 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 5 (6)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 6 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4) | 10 (11)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (8) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (13) | 29 (36)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days